CLINICAL TRIAL: NCT00439127
Title: Is the Thyroglobulin Measurement Under Thyroxine of Prognostic Value Before rhTSH-Aided Radioiodine Ablation in Differentiated Thyroid Carcinoma?
Brief Title: OnT4-Thyroglobulin Assay Before rhTSH-Aided Radioiodine Ablation
Status: Completed | Type: Observational
Sponsor: Oncology Institute of Southern Switzerland (Other)
Other Study IDs: IOSI-MN-1-07
Record Dates: First submitted 2007-02-22; First posted 2007-02-23 (Estimated); Last update posted 2007-02-28 (Estimated); Status verified 2007-02

CONDITIONS: Differentiated Thyroid Carcinoma
Keywords: thyroglobulin; thyroid carcinoma; tumour marker; radioiodine; recombinant human TSH
MeSH Terms: conditions — Thyroid Neoplasms

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
Thyroidectomy followed by administration of large activities of 131-iodine (131I) is the treatment of choice for differentiated thyroid carcinoma (DTC). The serum thyroglobulin (Tg) measurement during hypothyroidism (offT4-Tg), just before radioiodine thyroid ablation, has proved to be effective for predicting persistent/recurrent disease. However, the Tg measurement cannot be used as a corresponding value for preablative offT4-Tg when rhTSH is used as stimulous before treatment. The present study was undertaken to evaluate if post-thyroidectomy Tg values, measured before rhTSH-stimulation and radioiodine administration, is of prognostic value in patients affected by DTC. We enrolled 28 patients with DTC and submitted to total thyroidectomy. Thyroxine (T4) treatment was started just after surgery to suppress TSH levels. Six to nine weeks later Tg levels were measured both basally (onT4-Tg) and after rhTSH (rhTSH-Tg) stimulation. Subsequently, T4 was stopped and serum Tg measured (offT4-Tg) just before 3700 MBq of 131I-iodide administration. A post-treatment whole body scan (PT-WBS) was performed and neck radioiodine uptake (RAIU) measured. A significant relationship was found between onT4-Tg and both rhTSH-Tg and offT4-Tg. The onT4-Tg levels of 0.2 ng/mL or higher predicted PT-WBS results with a 100% negative and 43% positive predictive values, respectively. Additionally onT4-Tg levels of 0.9 ng/mL or more predicts 12-months recurrences with 100% negative and 60% positive predictive value. In comparison, 1.0 ng/mL or higher offT4-Tg values predicted PT-WBS results and 12-months restaging with 94% and 100% negative and 45% and 27% positive predictive value, respectively. Basing on our data we conclude that preablative onT4-Tg may be of value as prognostic marker when rhTSH-aided radioiodine ablation is done. Additionally, the role of preblative onT4-Tg measurement as a yard-stick for radioiodine ablation should be further evaluate.

DETAILED DESCRIPTION:
Introduction Total (or near-total) thyroidectomy followed by TSH-stimulated administration of large activities of 131-iodine (131I) is the treatment of choice for DTC [1-3]. The serum thyroglobulin (Tg) measurement during hypothyroidism, just before radioiodine thyroid ablation, has proved to be effective for predicting persistent/recurrent disease [4-8]. Recently recombinant human TSH (rhTSH) showed to be safely employed instead of thyroxine (T4) withdrawal (offT4) to prepare patients for radioiodine ablation [9-10]. However, the Tg level are measured 48 hours after radioiodine administration when rhTSH is used as stimulation [11]. Consequently, due to the radioiodine-induced thyroid cells damage and Tg release, the Tg measurement would not have reliable predictive value in patients treated by rhTSH stimulation [12]. The present study was undertaken to evaluate if preablativeTg measurement under T4 treatment is of prognostic value and serves as surrogate marker of offT4-stimulated preablative Tg.

Patients and methods

Patients selection We retrospectively enrolled 28 consecutive patients affected by histologically proven DTC (23 papillary, 5 follicular) submitted to total thyroidectomy and central compartment lymph-node dissection. Thyroxine (T4) treatment was started immediately after surgery to suppress TSH levels. Six to nine weeks later Tg levels were measured both basally (onT4-Tg) and after rhTSH (rhTSH-Tg) stimulation as previously described [13]. Subsequently, T4 was stopped for 4 weeks and serum Tg measured (offT4-Tg) just before 3700 MBq of 131I-iodide administration. A post-treatment whole body scan (PT-WBS) with radioiodine uptake (RAIU) calculation was performed according to a previously described protocol [1]. All non physiologic iodine uptake areas out of the thyroid bed were considered as positive findings [14, 15]. Patients with positive PT-WBS underwent specific treatment and personalized follow-up. Patients with negative PT-WBS immediately restarted T4 suppressive treatment. Final restaging was performed in all patients 12 months after the last treatment by neck ultrasound, onT4-Tg assay and both offT4-diagnostic WBS (DgWBS) and Tg assay (4 weeks T4 withdrawal; required TSH>30 mUI/L). Clinical and pathological characteristics of selected patients were summarized in the Table 1.

Serum Tg assay and screening for interferences Serum Tg was assayed in duplicate by a specific high-sensitive IRMA assay (DYNOtest® Tg-plus, BRAHMS Diagnostica GmbH, Berlin, Germany) according to the producer' instructions. This method provided a sensitivity of 0.05 ng/mL and a functional sensitivity of 0.2 ng/mL [16, 17]. As previously published, preablative offT4 serum Tg values above 4.5 ng/mL and 3.2 ng/mL were considered as positive with respect to PT-WBS and 12 months restaging results, respectively [8]. Otherwise, offT4-Tg values higher than 0.2 ng/ml measured 12 months after thyroid ablation were considered positive for persisting/relapsing disease. [18, 19]. The presence of anti-thyroglobulin antibodies (AbTg) was screened by a specific radioimmunoassay (DYNOtest® anti-TGn, BRAHMS Diagnostica GmbH, Berlin, Germany) and by recovery test with a specific Tg-recovery buffer provided by the producer. Sera showing AbTg levels more than 60 U/mL and/or recover less than 80% or more than 120% were excluded from the study. Quality control was ensured by assaying two levels of control sera in each series, by re-assessing all sera showing a coefficient of variation exceeding 10% and by a bimonthly partecipation in the European inter-laboratory control OncocheckTM.

Statistics Quantitative data are expressed as mean ± SD. Differences between groups were assessed by two-tailed unpaired t-test. The relationship between variables was assessed by linear regression analysis. In order to allow statistical analysis the value of undetectable serum Tg expressed as < 0.2 ng/nL was arbitrarily changed in 0.10 ng/mL. Statistical significance was defined by a p-value < 0.05.

Ethics All diagnostic and therapeutic procedures were performed according to the regulations of the local ethics committee. Informed consensus was obtained from each patient.

Results The overall results are summarized in the Table I. Relationship Between Post-surgery onT4-Tg, rhTSH-Tg and offT4-Tg A significant positive relationship was found between onT4-Tg and both rhTSH-Tg (p<.0001) and offT4-Tg (p<0.0001) (Figure 1, A-B-C) as well as between rhTSH and offT4-stimulated Tg (p<.0001).

Relationship Between Post-surgery Serum Tg and Thyroid Remnant Radioiodine Uptake (RAIU) Among 22 patients showing no DTC metastasis on PT-WBS the serum distribution of onT4-Tg, rhTSH-Tg and offT4-Tg was 0.342±0.402; 0.664±0.803 and 1.195±1.485 ng/mL respectively. Both rhTSH and offT4-stimulated Tg levels were related to RAIU (p <.05 and <.005, respectively) while no significant relationship was found between RAIU and onT4-Tg levels (Figure 1, D-E-F).

Relationship Between Post-surgery Serum Tg and PT-WBS results The patients with positive PT-WBS showed higher onT4-Tg (0.617±0.445 vs 0.341±0.402 ng/mL), rhTSH-Tg (2.150±1.249 vs 0.664±0.803 ng/mL) and offT4-Tg (4.417±2.136 vs 1.195±1.485 ng/mL) levels as compared with patients with negative scan. Among 14 patients with undetectable onT4-Tg (i.e. ≤0.2 ng/mL) none had positive PT-WBS neither recurrences at 12-months restaging. Additionally, none of these patients showed stimulated Tg values more than 0.4 ng/mL and 1.0 ng/mL after rhTSH stimulation and T4 withdrawal, respectively. Viceversa, among 14 patients with onT4-Tg levels more than 0.2 ng/mL, 6 had positive PT-WBS (onT4-Tg: 0.3 to 1.4 ng/mL) and 3 showed DTC recurrences at 12 months restaging (onT4-Tg: 0.9 to 1.7 ng/mL). Consequently, the onT4-Tg levels predicts PT-WBS results with a 100% negative and 43% positive predictive values, respectively. Additionally onT4-Tg levels of 0.9 ng/mL or more predicts 12-months recurrences with 100% negative and 60% positive predictive value. In comparison, 1.0 ng/mL or higher offT4-Tg values predicted PT-WBS results and 12-months restaging with 94% and 100% negative and 45% and 27% positive predictive value, respectively.

Discussion Many reports indicate the usefulness of Tg concentration measurement before radioiodine treatment to early detection of DTC relapse or metastasis [4-8, 20, 21]. Three factors determine Tg concentration in most clinical situations: thyroid cell mass, thyroid cell damage and activation of TSH receptors [22]. When Tg is measured before radioiodine ablation the effects of surgical damage are generally vanished and endogenous TSH levels are increased in all patients: consequently the thyroid remnant mass is the major determinant of the serum Tg concentrations [23]. However, the rhTSH-stimulated Tg cannot be used instead of preablative offT4-Tg when rhTSH is employed to prepare radioiodine ablation [12]. Therefore we evaluated the role of post-surgery onT4-Tg as surrogate prognostic marker. We choiced to suppress TSH levels in order to normalize the effect of TSH stimulation on thyroid remnants. Clearly, the TSH suppression reduced Tg levels: however, the high-sensitive Tg assays provide a good distinction between the lower limit of the euthyroid reference range and the functional sensitivity limit detecting small amounts of thyroid tissue even in the TSH-suppressed state (22, 23). We showed a significant positive relationship between post-surgery Tg measured during T4 treatment and after TSH stimulation. No relationship was found between RAIU (i.e. expression of remnant mass) and onT4-Tg, probably due the clustering of all Tg levels lower than 0.2 ng/mL (see statistics paragraph). However, undetectable onT4-Tg after surgery identifies patients free of metastasis at PT-WBS and without late recurreces during early 12-months follow-up. None of these patients showed a significant increase in both rhTSH and offT4-stimulated Tg before radioiodine ablation. This seems to indicate that the relationship between Tg expression and thyroid tissue mass is manteined even in TSH suppression state: Therefore undetectable serum onT4-Tg really identifies patients without significant thyroid tissue amount as well as stimulated Tg. All patients performed extracapsular total thyroidectomy in a dedicated thyroid surgery unit and the thyroid remnant, expressed as RAIU, was lower in our series than in others. This means that our data cannot directly translated to patients treated by more limited surgery. Globally, basing on our data we conclude that preablative onT4-Tg may be of value as prognostic marker when rhTSH-aided radioiodine ablation is done. Additionally, the role of preblative onT4-Tg measurement as a yard-stick for radioiodine ablation should be further evaluate.

References

1. Schlumberger MJ. Medical progress: papillary and follicular thyroid carcinoma. N Engl J Med 1998; 338: 297-306.
2. Pacini F. Follow-up of differentiate thyroid cancer. Eur J Nucl Med 2002; 29(S2): 492-6.
3. Klain M, Richard M, Leboulleux S et al. Radioiodine therapy for papillary and follicular thyroid carcinoma. Eur J Nucl Med 2002; 29(S2): S479-85.
4. Ronga G, Filesi M, Ventroni G et al. Value of the first serum thyroglobulin level after total thyroidectomy for the diagnosis of metastasis from differentiated thyroid carcinoma. Eur J Nucl Med 1999; 26(11): 1448-52.
5. Grünwald F, Menzel C, Fimmers R et al. Prognostic value of thyroglobulin after thyroidectomy before ablative radioiodine therapy in thyroid cancer. J Nucl Med 1996; 37(12): 1962-4.
6. Lin JD, Huang MJ, Hsu BR, Chao TC, Hsueh C, Liu FH et al. Significance of postoperative serum thyroglobulin levels in patients with papillary and follicular thyroid carcinomas. J Surg Oncol 2002; 80: 45-51.
7. Kim TY, Kim WB, Kim ES, Ryu JS, Yeo JS, Kim SC et al. Serum thyroglobulin levels at the time of 131I remnant ablation just after thyroidectomy are useful for early prediction of clinical recurrence in low-risk patients with differentiated thyroid carcinoma. J Clin Endocrinol Metab 2005; 90: 1440-5.
8. Giovanella L, Ceriani L, Ghelfo A, Keller F. Thyroglobulin assay 4 weeks after thyroidectomy predicts outcome in low-risk papillary thyroid carcinoma.Clin Chem Lab Med 2005;43: 843-7.
9. Barbaro D, Boni G, Meucci G, Simi U, Lapi P, Orsini P et al. Recombinant human thyroid-stimulating hormone is effective for radioiodine ablation of post-surgical thyroid remnants. Nucl Med Commun. 2006; 27(8):627-32.
10. Pacini F, Ladenson PW, Schlumberger M, Driedger A, Luster M, Kloos RT et al. Radioiodine ablation of thyroid remnants after preparation with recombinant human thyrotropin in differentiated thyroid carcinoma: results of an international, randomized, controlled study. J Clin Endocrinol Metab. 2006; 91: 926-32.
11. Robbins RJ, Svrivastava S, Shaha A, Ghossein R, Larson SM, Fleischer M et al. Factors influencing the basal and recombinant human thyrotropin-stimulated serum thyroglobulin in patients with metastatic thyroid carcinoma. J Clin Endocrinol Metab. 2004; 89: 6010-6.
12. Taieb D, Lussato D, Guedj E, Roux F, Mundler O. Early sequential changes in serum thyroglobulin after radioiodine ablation for thyroid cancer: possible clinical implications for recombinant human thyrotropin-aided therapy. Thyroid 2006; 16: 177-9.
13. Mazzaferri E, Robbins RJ, Spencer CA, Braverman LE, Pacini F, Wartofsky L et al. A consensus report of the role of serum thyroglobulin as a monitoring method for low-risk patients with papillary thyroid carcinoma. J Clin Endocrinol Metab 2003; 88: 1433-41.
14. Giovanella L, Ceriani L, Ghelfo A, Keller F, Sacchi A, Maffioli M et al. Thyroglobulin assay during thyroxine treatment in low-risk differentiated thyroid cancer management: comparison with recombinant human thyrotropin-stimulated assay and imaging procedures. Clin Chem Lab Med 2006; 44:248-52.
15. Reiners C, Luster M, Lassman M. Clinical experience with recombinant human thyroid-stimulating hormone (rhTSH): whole-body scanning with iodine-131. J Endocrinol Invest 1999; 22(S11):17-24.
16. Giovanella L, Ceriani. High-sensitivity human thyroglobulin (hTG) immunoradiometric assay in the follow-up of patients with differentiated thyroid carcinoma. Clin Chem Lab Med 2002; 40(5): 480-4.
17. Morghentaler NG, Froelich J, Rendl J, Willnich M, Alonso C, Bergmann A et al. Technical evaluation of a new immunoradiometric and a new immunoluminometric assay for thyroglobulin. Clin Chem 2002; 48(7): 1077-83.
18. Iervasi A, Iervasi G, Carpi A, Zucchelli GC. Serum thyroglobulin measurement: clinical background and main methodological aspects with clinical impact. Biomed Pharmacother. 2006; 60: 414-24
19. Sahlmann CO, Schreivogel I, Angerstein C et al. Clinical evaluation of a new thyroglobulin immunoradiometric assay in the follow-up of differentiated thyroid carcinoma. Nuklearmedizin 2003; 42: 71-7.
20. Makarewicz J, Adamczewski Z, Knapska-Kucharska M, Lewinski A. Evaluation of the diagnostic value of first thyroglobulin determination in detecting metastases after differentiated thyroid carcinoma surgery. Exp Clin Endocrinol Diabetes 2006; 114: 485-9.
21. de Rosario PW, Guinaraes VC, Maia FF, Fagundes TA, Purisch S, Padrao EL et al. Thyroglobulin before ablation and correlation with posttreatment scanning. Laryngoscope 2005; 115: 264-7.
22. Spencer CA, LoPresti JS, Fatemi S, Nicoloff JT. Detection of residual and recurrent differentiated thyroid carcinoma by serum thyroglobulin measurement. Thyroid 1999; 9: 435-41.
23. Wunderlich G, Zophel K, Crook L, Smith S, Smith BR, Franke WG. A high-sensitivity enzyme-linked immunosorbent assay for serum thyroglobulin. Thyroid 2001; 11: 819-24.

ELIGIBILITY:
Inclusion Criteria:

* Hiostologically proved DTC (M0)

Exclusion Criteria:

* Preoperative metastasis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 28
Dates: Start 2005-01; Study Completion 2007-01

CONTACTS AND LOCATIONS:
Overall Officials: Luca Giovanella, MD, Principal Investigator — Oncology Institute of Southern Switzerland